CLINICAL TRIAL: NCT03664765
Title: Novel Treatment of Sleep Apnea by Upper Airway and Respiratory Muscle Training
Brief Title: Novel by Upper Airway Respiratory Muscle Training to Treat OSA in Chronic SCI
Acronym: NOURMT-OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2885-P
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: OSA; SCI/D; Upper Airway Exercise
Keywords: OSA; SCI/D; RMT; Upper airway exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot trial to assess the feasibility of using combined oropharyngeal and respiratory muscle training versus sham training on OSA in patients with chronic SCI/D
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized and blinded to the intervention arm (upper airway and respiratory muscle training arm) versus sham arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention exercise arm (Active Comparator): daily oropharyngeal and respiratory muscle exercises
  Interventions: Other: UA and RMT
- Control arm (Sham Comparator): Daily sham exercises
  Interventions: Other: Sham exercise

INTERVENTIONS:
Other: UA and RMT — daily oropharyngeal and respiratory muscle exercises
  Arms: Intervention exercise arm
Other: Sham exercise — Daily sham exercises
  Arms: Control arm

SUMMARY:
It is estimated that spinal cord injury (SCI) affects approximately 12,000 new individuals every year in the United States, with the majority are cervical and/or upper thoracic injuries. Despite this high prevalence of obstructive sleep apnea (OSA) in chronic SCI population minority of patients are treated and are adherent to standard therapy (CPAP). This proposal addresses a new therapeutic intervention for OSA in SCI. The investigators hypothesized that combined oropharyngeal and respiratory muscle exercises improve respiratory symptoms and alleviate OSA in patients with chronic SCI. The investigators will perform a pilot randomized, sham-controlled study to examine the impact of combined daily exercises (~30 min) for 1 and 3 months durations among Veterans with SCI. The investigators believe that this novel approach to treating OSA and will yield significant new knowledge that improves the health and quality of life of these patients.

DETAILED DESCRIPTION:
In recent years, the investigators and others have discovered that spinal cord injury/disease (SCI/D) is associated with significant increase in the sleep-disordered breathing (SDB) prevalence. Nearly 80% of patients with SCI/D including Veterans suffer from SDB after six months of injury (majority of them 70-80% are obstructive apneas and hypopneas-OSA). However, most patients SCI/D do not tolerate standard SDB treatment (continuous positive airway pressure-CPAP) leading to lack of compliance. Therefore, identifying other therapies is important for this common condition that is linked to poor outcome in the general population (heart disease, stroke, hypertension and poor cognition). It has been reported in sleep apnea able-bodied patients that oropharyngeal muscle exercises for 3 months using speech pathology techniques improve the severity of SDB. Furthermore, previous studies showed respiratory muscle training (RMT) is effective for increasing respiratory muscle strength in people with cervical SCI. However, the effect of combined oropharyngeal and RMT on OSA in patients with SCI is unknown.

The purpose of this application is to identify new therapeutic interventions for OSA treatment in Veterans with SCI/D. This application proposes for a pilot study to randomizing 30 Veterans with SCI/D and OSA to receive 3 months of daily (30 minutes) treatment with a validated set of oropharyngeal and RMT (intervention arm) versus sham therapy (control arm). There will be three specific aims to address the following hypotheses:

Specific Aim (1): To test recruitment rate and feasibility of a pilot intervention that includes combined oropharyngeal and RMT versus sham treatment in individuals with SCI/D.

Specific Aim (2): To test the acceptability and usability of combined oropharyngeal and RMT in individuals with SCI/D.

Specific Aim (3): To determine the effect size estimates for clinical endpoints and their associated variability at the end of treatment to calculate an appropriate sample size for an adequately powered clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic SCI/D (>6 months post-injury)
* American Spinal Injury Association (ASIA) classification A-D who have evidence of OSA

  * excluding those with no evidence of a neurologic deficit based on ASIA classification
* Specifically, the study will target those with SCI/D and OSA who would like alternative treatment options or to have a lower PAP pressure, if they refused, or did not tolerate PAP treatment

Exclusion Criteria:

* Receiving continuous mechanical ventilation

  * except PAP therapy which is considered usual treatment for SDB)
* Severe congestive heart failure with ejection fraction <35%
* Recent health event that may affect sleep

  * stroke
  * acute myocardial infarction
  * recent surgery
  * hospitalization
* Alcohol or substance abuse (<90 days sobriety)
* Self-described as too ill to engage in study procedures
* Unable to provide self-consent for participation
* Central sleep apnea (CSA) defined as central apnea/hypopnea index >50% of the AHI

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulghani Sankari, MD PhD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publications from research will be made available to the public through the national Library of Medicine PubMed within one year after the date of publication. Final data sets underlying all publications resulting form the proposed research will be shared outside if the following criteria is met: A limited Dataset will be created and shared pursuant to Data Use Agreement (DUA) appropriately limiting use for dataset and prohibiting the recipient from identifying or re-identifying any individuals whose data are included in the dataset.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of the publication

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to the primary site at John D. Dingell VA Medical Center.
Pre-assignment Details: Of 188 screened, 29 participants were enrolled. Of the 29 enrolled, 24 started the study protocol.
Period: Overall Study
Arm/Group | Intervention Exercise Arm | Control Arm
Started | 12 | 12
Completed | 8 | 10
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Exercise Arm | Control Arm | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.0) | 64.8 (7.7) | 65.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 8 | 4 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Feasibility-Number of Participants Who Complete the Three-month Protocol
Description: Assess the feasibility of completing intervention arm (upper airway and respiratory muscle training arm) verses sham arm.
Time Frame: 3 months
Population: This measures the number of randomized participants who stayed active in the study long enough to complete the three month protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Exercise Arm | Control Arm
Number analyzed (Participants) | 12 | 12
Participants | 8 | 10

2. Primary Outcome: Recruitment
Description: Assess the recruitment rate of the study
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Groups:
- Recruited Portion of Eligible Pool: This is the portion of the screened individuals who were found to be eligible that agreed to enroll in the study.
Arm/Group | Recruited Portion of Eligible Pool
Number analyzed (Participants) | 80
Participants | 29

ADVERSE EVENTS:
Time Frame: Adverse event information was collected during the duration of time that the participants were performing exercises (3 months).
Arm/Group | Intervention Exercise Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
- The sample size is small and the majority are males, therefore findings from this study may not be applicable to the general population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT03664765/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03664765/ICF_001.pdf